CLINICAL TRIAL: NCT05991011
Title: Moving While Thinking or Thinking While Moving? Comparison of the Cognitive, Dual-task and Physical Effects of 6 Programs With Older Adults
Brief Title: Comparison of the Cognitive, Dual-task and Physical Effects of 6 Programs With Older Adults
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Alexandra Perrot (Other)
Collaborators: Université Paris Cité (Other)
Responsible Party: Sponsor-Investigator, Alexandra Perrot, Principal Investigator, Université Paris-Saclay
Organization: Université Paris-Saclay (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: UParis-Saclay
Record Dates: First submitted 2023-07-13; First posted 2023-08-14 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Physical Fitness; Cognitive Function
Keywords: exergames; combined training; cognitive function; dual task; older adults; video games; physical activity
MeSH Terms: conditions — Motor Activity | interventions — Off-Road Motor Vehicles

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- I2WE (Immersive and interactive wall exergames) (Experimental)
  Interventions: Other: Immersive and Interactive Wall Exergames
- 2CMA (Complex Cognitive and Motor Activities) (Experimental)
  Interventions: Other: Complex Cognitive and Motor Activities program
- EXER (Experimental)
  Interventions: Other: exergames program
- VG (video games) (Active Comparator)
  Interventions: Other: video games program
- BIKE (bike) (Active Comparator)
  Interventions: Other: Bike
- VG-bike (Video games + bike) (Active Comparator)
  Interventions: Other: Video games + bike
- CON (control group) (No Intervention)

INTERVENTIONS:
Other: Immersive and Interactive Wall Exergames — This intervention will be performed using the Neo One device. It was chosen because of the variety and quality of the games offered which are accessible to older people. The target intensity of core workout will be moderate. Five to 7 five-minutes games will be selected from 19 games. A variety of materials will be used (e.g., basketball, rugby, handball ball, balloon, chair, hoop, rhythm ladder, tennis racket). The games will be made more complex by selecting difficulty settings (easy, normal, hard) and by adding extra exercises to add cooperative and/or oppositional situations to the games where they are not initially implemented and to increase the physical and/or motor complexity. Interventions will last 12 weeks, with 2 sessions of 1-h per week (24 h in total). The sessions will consist in 10 minutes of warmup, 45 minutes of the main session using the Neo One device and 5 minutes of cooldown with full body stretching exercises, in groups of 4 participants.
  Arms: I2WE (Immersive and interactive wall exergames)
Other: Complex Cognitive and Motor Activities program — The intervention will last 12 weeks, with 2 sessions of 1-h per week (24 h in total). The sessions will consist in 10 minutes of warmup, 45 minutes of the main sessions involving cooperation and opposition exercises inspired by team sports (basketball, volleyball, rugby) and individual sports (boxing, weight training), and 5 minutes of cooldown with full body stretching exercises, in groups of 6 participants. The target intensity of body workout will be moderate. The first part will be focused on endurance and the second on muscle strengthening and coordination work in the form of circuit training. A variety of equipment will be used (e.g., tennis balls, basketballs, volleyballs, rugby balls, balloons, elastics, chairs, blocks). The number of partners and/or opponents will be changed regularly.
  Arms: 2CMA (Complex Cognitive and Motor Activities)
Other: exergames program — The intervention will last 12 weeks, with 2 sessions of 1-h per week (24 h in total). The sessions will be performed using the Nintendo Switch device, physically active (standing). The sessions will consist in 10 minutes of warmup, 45 minutes of the main session using the Nintendo Switch device and 5 minutes of cooldown with full body stretching exercises, in groups of 4 participants. The games (Fitness Boxing 2, Switch Sport, Just Dance 2020, 2021, 2023, Let's Get Fit, Mario and Sonic at the Olympic Games Tokyo 2020, Instant Sport, Ring Fit, Zumba Burn It Up!) will be carried out in the form of circuit training, in pairs or groups of 4. The games will be made more complex by selecting difficulty settings (easy, normal, hard) and by adding extra exercises to add cooperative and/or oppositional situations to the games where they are not initially implemented and to increase the physical and/or motor complexity.
  Arms: EXER
Other: video games program — The intervention will last 12 weeks, with 2 sessions of 1-h per week (24 h in total). The sessions will be performed using the Nintendo Switch device, while being inactive (sitting). The sessions will consist in one-hour single and multi-players games, using the Nintendo Switch device, in groups of 6 participants.
  Arms: VG (video games)
Other: Bike — The intervention will last 12 weeks, with 2 sessions of 1-h per week (24 h in total). In this active comparator intervention, the sessions will consist in 10 minutes of warmup, 45 minutes of the main sessions involving riding a stationary bike at about 50% of Heart Rate Reserve, and 5 minutes of cooldown with full body stretching exercises, in groups of 6 participants.
  Arms: BIKE (bike)
Other: Video games + bike — The intervention will last 12 weeks, with 2 sessions of 1-h per week (24 h in total). In this experimental arm, the sessions will consist in 10 minutes of warmup, 45 minutes of the main sessions involving riding a stationary bike (like BIKE program at about 50% of Heart Rate Reserve) and at the same time playing on a Nintendo Switch (like VG program), and 5 minutes of cooldown with full body stretching exercises, in groups of 6 participants.
  Arms: VG-bike (Video games + bike)

SUMMARY:
While the association of physical and/or motor and/or cognitive components with training can generate synergistic effects and thus create an efficient cognitive enrichment program, very few studies have focused on finding an optimal combined program for older adults. According to the model of Herold and his colleagues, there are two modalities of simultaneous combined training: Thinking While Moving (TwM), when the additional cognitive task is not linked to the motor task, and Moving While Thinking (MwT), when the cognitive task is integrated into the motor task. They assume the latter approach is the most promising for improving cognitive reserve. Nevertheless, to the investigators' knowledge, only one study has compared these two modalities in older adults and none has broadened the question by comparing several MwT trainings.

The goal of this interventional study will be to compare the cognitive, dual-task, and physical effects of 6 physical and/or cognitive programs in healthy but inactive older adults. The main questions it will aims to answer are:

* Will the Moving While Thinking and Thinking While Moving programs have the same effects?
* If they have different effects, which will be the best way to improve cognitive, dual-task, and physical functions? The study is being set up between 2023 and 2025 to compare the cognitive, dual- ask and physical effects of 6 programs (3 months, 2 sessions of 1 hour per week). Three experimental MwT programs will be studied: Immersive and interactive wall exergames (I2WE), Complex Cognitive and Motor Activities (2CMA), and exergames with Switch (EXER). They will be compared to an experimental TwM program of stationary bike simultaneous to the Switch (Video games + bike) and 2 control programs: inactive video games (VG) and stationary bike (BIKE). A control group (CON) will be also created.

Cognitive, dual-task, and physical pre-tests (before the program), post-tests (after the program), and retention tests (3 months after the end of the program) will be realized to evaluate the effects of the programs.

DETAILED DESCRIPTION:
All subjects must give their informed consent for inclusion before they participate in the study. The study will be conducted in accordance with the Declaration of Helsinki, and the protocol has been approved by the University Paris Saclay Ethics Committee of Research (N°462) who stated that a Protection of Persons Committee was not necessary. The sample size calculation was performed using G. Power. The investigators calculated a sample size sufficient to detect small effect sizes (η2 = .04). Therefore, f = 0.20, α = 0.05, p = 0.95, power = 0.95, were chosen to favor clinically significant effect sizes. To test the main hypotheses of the present study, 133 participants are required. To compensate for possible dropouts, 35 more participants will be included. The 7 groups will be composed of 24 participants each, for a total of 168 participants.

The training interventions will be carried out in different places and at different times:

* Montreuil for I2WE and 2CMA (February to May 2023)
* Créteil for EXER (September to December 2023)
* Paris for BIKE and VG-BIKE (February to May 2024)
* Orsay for VG (September to December 2023). Pre- and post-tests will be carried out before and after the training period to evaluate the cognitive, DT, and physical benefits of each program, and retention tests 3 months after the end of the program.

Statistical analysis plan: Data will be analyzed with JASP software. The statistical analysis will allow us to determine the effects of the 7 different groups on the cognitive, DT, and physical functions. The analysis will include only subjects who completed all the pre- and post-tests. Data from the pre-tests, post-tests, and retention tests will be presented using descriptive statistics (mean, standard deviation) to describe the participants' characteristics and performances on assessments. Before performing the inferential statistical tests, all relevant hypotheses will be tested, and if they are met, statistical analysis will be conducted. For primary and secondary measures, repeated ANOVA will be used to test the interaction between pre-test, post-test, retention test x training groups. If a significant interaction is found, a Bonferroni post-hoc test will be performed. Effects sizes will be calculated to study the power of the results.

ELIGIBILITY:
Inclusion Criteria:

* be over 60 years old
* have a MMSE score above 27
* engage in less than 2.5 hours of physical activity per week assessed by the QAPPA
* score 3 or higher on a subjective health Likert-scale (1= very poor to 5= very good)
* be retired
* have no major pathology
* have normal or corrected vision and hearing
* have no difficulty bending or using their shoulders
* do not frequently play video games or exergames
* present a medical certificate not contraindicating physical activity).

Exclusion Criteria:

-

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 168 (Estimated)
Dates: Start 2023-02-13 (Actual); Primary Completion 2024-12-15 (Estimated); Study Completion 2025-05-15 (Estimated)

PRIMARY OUTCOMES:
Change Visuospatial memory | Within 1 week before the program, within 1 week after the program, and 3 months after the end of the program.
  Visuospatial memory will be evaluated with the Spatial Span Test, a subtest of the Weschler Memory Scale. In the first part, the participant reproduces in the same order a sequence of cubes designated by the examiner. In the second, the participant reproduces a sequence of movements in reverse order. The number of cubes increases progressively and determines the spatial span and the backward spatial span. For each level, the participant always performs 2 trials and scores 1 point for each successful trial. The test ends when 2 errors are made at the same level.
Change Flexibility | Within 1 week before the program, within 1 week after the program, and 3 months after the end of the program.
  Flexibility will be evaluated with the Trail Making Test. Part A consists in linking a series of increasing numbers from 1 to 25 by selecting the appropriate number. In part B, the participants connect 2 series of symbols in alternation: 1 of numbers and 1 of letters. This has to be done without lifting the pen from the paper and as quickly as possible. If mistakes are made, the examiner informs the participant, who has to correct them. Flexibility is highlighted specifically by analyzing the time difference in the result B-A, a purer measure of flexibility.
Change Inhibition with witty | Within 1 week before the program, within 1 week after the program, and 3 months after the end of the program.
  It will be performed with a set of eight semaphores which are equipped with a LED matrix. The participant will be standing, facing a specially designed rack with semaphores. They will have to turn off as fast as possible the lights that appear, according to the instructions given, and will have to move back their hand to the middle of their hips. The tests consist of 20 trials, each trial starts 1500ms after the previous response. The total time to complete the tests will be recorded in milliseconds. In part A, the participant will have to turn off the semaphores that were randomly lit up red. The others remained unenlightened. In part B, the participant will have to turn off the semaphores that were randomly lit up with the green letter O. The others lit up with other colors associated with a letter. In part C, the participant will have to turn off the semaphores randomly lit up with the green letter O. The others lit up in green are associated with another letter.
Change cognitive-cognitive Dual task | Within 1 week before the program, within 1 week after the program, and 3 months after the end of the program.
  To evaluate the cognitive-cognitive Dual Task capacity, the cognitive tasks will be first realized separately as a single task, and then concomitantly. For the Sound counting task, the participant will have to count in their mind the number of high-pitched sounds among low-pitched sounds that they heard, for 2 minutes. At the end of the 2 minutes, the participant will have to give the number of high-pitched sounds counted. The percentage between the number given by the participant and the correct number will be calculated. For the Go no Go Test, the participant will have to press a key as quickly as possible when they see the "X" symbol and not press when they see the "+" symbol, for 2 minutes. The reaction time, the number of correct answers, and errors will be recorded.
Change physical-cognitive Dual Task | Within 1 week before the program, within 1 week after the program, and 3 months after the end of the program.
  To evaluate the physical-cognitive Dual Task capacity, the cognitive and the physical task will be first realized separately as a single task, and then concomitantly. For the Operation counting task, the participant will subtract 7 from a starting number (e.g., 286) as many times as possible for one minute. The number of correct answers, as well as errors, will be recorded. For the STEP test, the participant will do as many repetitions as possible, going up and down a step, one foot after the other, for 2 minutes.

SECONDARY OUTCOMES:
Upper body strength change | Within 1 week before the program, within 1 week after the program, and 3 months after the end of the program.
  Upper body strength will be evaluated with the Chair-stand test. The participant will have to stand and sit up as many times as possible in 30 seconds. The arms will be crossed on the chest, the feet still on the ground. The number of chair-stand will be recorded.
Lower body flexibility change | Within 1 week before the program, within 1 week after the program, and 3 months after the end of the program.
  Lower body flexibility will be evaluated with the Chair-sit-and-reach test. Sitting on the edge of a chair, one leg straight, the other bent, the participant will have to bring their hand as close as possible to the foot of the straight leg. The number of centimeters between the hand and the foot will be measured. The values are negative if the fingers of the hand extended beyond the toes.
Dynamical balance change | Within 1 week before the program, within 1 week after the program, and 3 months after the end of the program.
  The dynamical balance will be evaluated with the TUG test. The participant will have to get up from a chair, walk around a block located in front of them, 3 meters away, and sit down again as quickly as possible. The time to complete this course will be recorded.
Upper body flexibility change | Within 1 week before the program, within 1 week after the program, and 3 months after the end of the program.
  Upper body flexibility will be evaluated with the Back-scratch test. The participant will have to bring their two hands as close together as possible (one hand reaching over the shoulder, palm against the back, the other reaching to the middle of the back, back of the hand against the back). The number of centimeters between both hands will be measured. The values are negative if the fingers of the two hands crossed.
Endurance change | Within 1 week before the program, within 1 week after the program, and 3 months after the end of the program.
  Endurance will be evaluated with the 6-min walking test. The participant will have to walk as far as possible, in 30-meter round trips, for 6 minutes. The distance will be recorded, as well as the heart rate to determine the intensity of the effort.
Upper body strength change | Within 1 week before the program, within 1 week after the program, and 3 months after the end of the program.
  Upper body strength will be evaluated with the Handgrip test. The participant will have to squeeze a dynamometer with maximum isometric effort, which has to be maintained for about 5 seconds. The force created, measured in kilograms, will be recorded for both arms.
Upper body strength 2 change | Within 1 week before the program, within 1 week after the program, and 3 months after the end of the program.
  Upper body strength will be also evaluated with the Seated Medicine Ball Throw test. Sitting in a chair, back against the back of the chair, feet flat on the floor, the subject will have to throw a 3kg medicine ball as far as possible with both hands, starting from the chest. The distance between the subject and the medicine ball will be recorded.
Coordination change | Within 1 week before the program, within 1 week after the program, and 3 months after the end of the program.
  Coordination will be evaluated with the Rhythm Ladder test. The participant will have to cross as quickly as possible, and with as few mistakes as possible, a 3-meter rhythmic ladder placed on the ground. To cross the ladder, they will have to respect a sequence of foot movements: put two feet consecutively in the first square, then two feet consecutively on both sides of the same square, then put two feet in the next square, then outside, and so on. The time to complete the test and the number of errors will be recorded.

OTHER OUTCOMES:
Perceived pleasure | within 1 week after the program
  The French version of the Physical Activity Enjoyment Scale with a scale from completely disagree (1) to completely agree (7) will be used to evaluate the perceived pleasure. The score will be between 7 and 70. Higher scores mean a better outcome.
Feeling questionnaire | within 1 week after the program
  The feeling questionnaire will be completed at the end of the program. It will consist of 4 questions following a 5-point Likert-scale, concerning (a) the difficulty of the sessions, (b) their physical and (c) cognitive developments, and (d) the desire to continue a program of this type. The score will be between 1 and 5 for each element. Higher scores mean a better outcome
General Lifestyle change | Within 1 week before the program, within 1 week after the program, and 3 months after the end of the program.
  The General Lifestyle Questionnaire (GLQ) assesses 46 types of behaviors and activities practiced in the last 12 months. The GLQ assesses five dimensions of lifestyle: "physical," "cognitive," "social," "other leisure activities" and "sleep and consumption (food, tobacco and alcohol)." The GLQ scores are calculated according to the frequency of practice of each activity or behavior. For each item, participants will indicate the frequency on a 5-point Likert-scale scoring 1 = never, 2 = a few times in the last year, 3 = a few times per month, 4 = a few times per week, 5 = every day or almost every day, and 8 items use inverse scoring. The averages of the five dimensions will be calculated, as well as the overall mean.
Physical effort intensity | up to 12 weeks
  effort intensity will be evaluated at each season with a Polar Verity Sense heart rate monitor. The Heart Rate Reserve (HRR), the difference between the Maximum Theoretical Heart Rate (MTHR = 192 - 0.007 x age²) and the Resting Heart Rate (RHR), is used to calculate exercise intensity. For all sessions, the mean intensity was calculated [(Average Heart Rate - RHR)/HRR] x 100]
perceived physical effort intensity | up to 12 weeks
  perceived effort intensity will be evaluated with the modified Borg Scale, a Likert scale from 0 to 10, with 0 = complete rest and 10 = extremely strong).
perceived cognitive effort intensity | up to 12 weeks
  perceived cognitive effort intensity will be evaluated with a Likert scale from 0 to 10, with 0 = complete rest and 10 = extremely strong).

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra Perrot, Study Director — Université Paris-Saclay; Pauline Maillot, Study Director — Université Paris Cité
Locations (3):
- France (3):
  - Club seniors Kennedy, Créteil
  - Centre Sportif Arthur Ashe, Montreuil
  - UFR STAPS Paris Cité, Paris

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Borg GA. Psychophysical bases of perceived exertion. Med Sci Sports Exerc. 1982;14(5):377-81. PMID 7154893
- [Background] de Souto Barreto P. Construct and convergent validity and repeatability of the Questionnaire d'Activite Physique pour les Personnes Agees (QAPPA), a physical activity questionnaire for the elderly. Public Health. 2013 Sep;127(9):844-53. doi: 10.1016/j.puhe.2012.10.018. Epub 2012 Nov 10. PMID 23148890
- [Background] Eggenberger P, Schumacher V, Angst M, Theill N, de Bruin ED. Does multicomponent physical exercise with simultaneous cognitive training boost cognitive performance in older adults? A 6-month randomized controlled trial with a 1-year follow-up. Clin Interv Aging. 2015 Aug 17;10:1335-49. doi: 10.2147/CIA.S87732. eCollection 2015. PMID 26316729
- [Background] Folstein MF, Folstein SE, McHugh PR. "Mini-mental state". A practical method for grading the cognitive state of patients for the clinician. J Psychiatr Res. 1975 Nov;12(3):189-98. doi: 10.1016/0022-3956(75)90026-6. No abstract available. PMID 1202204
- [Background] Gellish RL, Goslin BR, Olson RE, McDonald A, Russi GD, Moudgil VK. Longitudinal modeling of the relationship between age and maximal heart rate. Med Sci Sports Exerc. 2007 May;39(5):822-9. doi: 10.1097/mss.0b013e31803349c6. PMID 17468581
- [Background] Herold F, Hamacher D, Schega L, Muller NG. Thinking While Moving or Moving While Thinking - Concepts of Motor-Cognitive Training for Cognitive Performance Enhancement. Front Aging Neurosci. 2018 Aug 6;10:228. doi: 10.3389/fnagi.2018.00228. eCollection 2018. PMID 30127732
- [Background] Kraft E. Cognitive function, physical activity, and aging: possible biological links and implications for multimodal interventions. Neuropsychol Dev Cogn B Aging Neuropsychol Cogn. 2012;19(1-2):248-63. doi: 10.1080/13825585.2011.645010. PMID 22313174